CLINICAL TRIAL: NCT01219777
Title: Phase I Evaluation of Intravenous Carboplatin With Weekly Paclitaxel and Bevacizumab in Patients Undergoing Neoadjuvant Chemotherapy for Epithelial Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Neoadjuvant Chemotherapy IV Carboplatin With Weekly Paclitaxel \Bevacizumab for Primary Ovarian
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ritu Salani (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ritu Salani, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09149; NCI-2012-00512 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2015-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: bevacizumab; paclitaxel; carboplatin; ovarian; cancer; fallopian tube; primary peritoneal
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Carboplatin; Bevacizumab; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Carboplatin (Experimental): AUC 5.0 or 6.0
  Interventions: Drug: carboplatin
- Bevacizumab (Experimental): 15 mg/kg
  Interventions: Drug: Bevacizumab
- Paclitaxel (Experimental): 60-80 mg/m2
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: carboplatin — Carboplatin AUC 5.0 or 6.0 will be administered on day 1 during cycle 1-3. Treatment cycle consists of 21 days duration.
  Other Names: Paraplatin®; CBDCA
  Arms: Carboplatin
Drug: Bevacizumab — Bevacizumab 15 mg/kg administered on Day 1 during cycle 1-3. Treatment cycle consists of 21 days duration.
  Other Names: Avastin
  Arms: Bevacizumab
Drug: Paclitaxel — 60-80 mg/m2 administered on Day 1, 8 & 15 during cycle 1-3. Treatment cycle consists of 21 days duration.
  Other Names: Taxol; Abraxane
  Arms: Paclitaxel

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of intravenous weekly paclitaxel given with intravenous carboplatin and bevacizumab in patients with epithelial ovarian, primary peritoneal, or fallopian tube carcinoma that are to receive neoadjuvant chemotherapy (prior to surgical cytoreduction). Patients will then undergo surgery which will allow an objective measure of response to the above regimen as well as assessment of surgical outcomes.

DETAILED DESCRIPTION:
Phase I study proposed to evaluate:

* Tolerability of IV regimen carboplatin, paclitaxel and bevacizumab in the neoadjuvant setting prior to surgery.
* Safety/Toxicity of IV regimen in this patient population
* Treatment is Carboplatin area under the concentration curve (AUC) 5, Bevacizumab 15mg/m2, and starting dose of paclitaxel of 60mg/m2 and will be escalated in intervals of 10mg/m2 to a maximum dose of 80mg/m2.
* Patients will receive cycles 1-3 of carboplatin, bevacizumab, and paclitaxel and then cycle 4 will be carboplatin and paclitaxel followed by surgical intervention within 6 weeks of cycle 4.
* Post surgical treatment per physician discretion

ELIGIBILITY:
Inclusion Criteria:

* histology,cytologically diagnosed epithelial ovarian, primary peritoneal or fallopian tube cancer
* FIGO (International Federation of Gynecology and Obstetrics stage III or IV disease
* GOG (Gynecologic Oncology Group) Performance Status 0,1,2
* No prior surgery for their malignancy
* Adequate bone marrow function
* Platelet count greater than or equal to 100,000
* Renal Function: Creatinine < 1.5 institutional upper limit normal
* Hepatic Function: Bilirubin less than 1.5 ULN (upper limit of normal)
* Hepatic Function: SGOT (serum glutamate oxaloacetate transaminase) and Alkaline Phosphate
* Neurologic Function: Neuropathy less than CTCAE (Common Toxicity Criteria for Adverse Effects)grade 1
* Coagulation Functions: INR<1.5 and PTT ,1.2 times the upper limit of normal
* Measurable disease

Exclusion Criteria:

* Previous cancer related surgery
* Received prior chemotherapy, immunotherapy, radiotherapy, hormonal therapy or biologic therapy for their ovarian, fallopian tube or primary peritoneal cancer.
* Borderline ovarian tumors, recurrent epithelial ovarian or primary peritoneal cancer or non-epithelial ovarian are not eligible.
* Other cancers within 5 years (other than non-melanoma skin cancer)
* Acute Hepatitis or end stage liver disease
* History of prior gastrointestinal perforation
* Evidence of abdominal free air not explained by paracentesis
* Sign or symptoms of gastrointestinal obstruction
* Active bleeding or pathologic conditions that carry high risk of bleeding
* CNS (Central Nervous System) disease
* Clinically Significant cardiovascular disease
* Known hypersensitivity to Chinese Hamster ovary cell products or other recombinant human or humanized antibodies
* Clinically significant proteinuria.
* Hypertensive crises or hypertensive encephalopathy
* History of hemoptysis
* Any non-study related invasive procedure within 28 days fo first date of bevacizumab
* GOG performance status 3 or 4
* Patients who are pregnant or nursing.
* Under the age of 18
* Received prior treatment of bevacizumab or any anti-VEGF (vascular endothelial growth factor) drug

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Salani, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from January to December 2011.
Pre-assignment Details: Patients with a histologically or cytologically confirmed EOC with radiographic evidence of advanced disease, consistent with FIGO stage IIIC or IV.
Groups:
- Carboplatin + Weekly Paclitaxel and Bevacizumab: * Chemotherapy Cycles 1-3: After study enrollment all patients will receive 3 cycles of carboplatin, weekly paclitaxel and bevacizumab. The cycles will be administered every 21 days.
  * Chemotherapy Cycle 4: Enrolled patients will receive carboplatin and paclitaxel without bevacizumab for cycle 4. Radiologic imaging will be obtained pretreatment and after cycle 4.
  * Surgery: After 4 cycles of chemotherapy patients will be evaluated for surgical exploration. Patients who complete treatment with neoadjuvant chemotherapy and are medically fit, will undergo maximal tumor cytoreduction. Surgery should be undertaken at least 28 days after the administration of bevacizumab.
  * Post-Surgical Chemotherapy: Following surgery, chemotherapy will be at the discretion of the treating physician and will not be part of the study outcomes. There currently is no standard therapy for patients with ovarian cancer after undergoing interval debulking, therefore, this will be at the discretion of
Period: Overall Study
Arm/Group | Carboplatin + Weekly Paclitaxel and Bevacizumab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: * Chemotherapy Cycles 1-3: All patients will receive 3 cycles of carboplatin, weekly paclitaxel and bevacizumab. Cycles will be administered every 21 days.
  * Chemotherapy Cycle 4: Patients will receive carboplatin and paclitaxel without bevacizumab for cycle 4. Radiologic imaging will be obtained pretreatment and after cycle 4.
  * Surgery: After 4 cycles of chemotherapy patients will be evaluated for surgical exploration. Patients who complete treatment with neoadjuvant chemotherapy and are medically fit, will undergo maximal tumor cytoreduction. Surgery should be undertaken at least 28 days after the administration of bevacizumab.
  * Post-Surgical Chemotherapy: Following surgery, chemotherapy will be at the discretion of the treating physician and will not be part of the study outcomes. There currently is no standard therapy for patients with ovarian cancer after undergoing interval debulking, therefore, this will be at the discretion of
Arm/Group | Arm I
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Tolerated Dose
Description: To determine the maximum tolerated dose of carboplatin AUC5 administered Day 1 Cycles 1-4, weekly paclitaxel 60-80mg/m2 administered on Day 1, 8,and 15 for 3 weeks cycles 1-4, bevacizumab 15mg/kg administered Day 1 Cycles 1-3 prior to surgical intervention.
Time Frame: Up to 6 months
Measure: Number; unit: mg/m^2
Groups:
- Arm I: * Chemotherapy Cycles 1-3: After study enrollment all patients will receive 3 cycles of carboplatin, weekly paclitaxel and bevacizumab. The cycles will be administered every 21 days.
  * Chemotherapy Cycle 4: Enrolled patients will receive carboplatin and paclitaxel without bevacizumab for cycle 4. Radiologic imaging will be obtained pretreatment and after cycle 4.
  * Surgery: After 4 cycles of chemotherapy patients will be evaluated for surgical exploration. Patients who complete treatment with neoadjuvant chemotherapy and are medically fit, will undergo maximal tumor cytoreduction. Surgery should be undertaken at least 28 days after the administration of bevacizumab.
  * Post-Surgical Chemotherapy: Following surgery, chemotherapy will be at the discretion of the treating physician and will not be part of the study outcomes. There currently is no standard therapy for patients with ovarian cancer after undergoing interval debulking, therefore, this will be at the discretion of
Arm/Group | Arm I
Number analyzed (Participants) | 9
mg/m^2 | 80

2. Secondary Outcome: Toxicity and Response Rates Based on Imaging and Surgical Outcomes
Description: Determine the safety/toxicity of this regimen in this patient population. Estimate the percent of patients undergoing successful cytoreductive surgery to optimal disease (<1 cm greatest tumor diameter) following neoadjuvant chemotherapy with carboplatin, paclitaxel and bevacizumab in patients with epithelial ovarian cancer, primary peritoneal cancer and fallopian tube cancer. Assess the 30 day morbidity and mortality following surgical intervention. To describe the response rate for patients treated with neoadjuvant carboplatin, weekly paclitaxel, and bevacizumab using RECIST and GCIG response criteria prior to surgical intervention. Response was determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Measure: Number; unit: patients
Arm/Group | Arm I
Number analyzed (Participants) | 9
patients
  Partial Responses | 9
  Dose Limiting Toxicities | 0
  Optimal debulking achieved | 9

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: The NCI Common Terminology Criteria for Adverse Events version 4.0 was used for toxicity assessment for patients.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=9)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Venous thromboembolic disease (Vascular disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes